CLINICAL TRIAL: NCT03891732
Title: The Use of MRI Prostate in Improving Detection of Significant Prostate Cancer in a Screening Population of Chinese Men With Elevated PSA
Brief Title: MRI Prostate for Chinese Men Being Screened for Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRE 2018.495
Record Dates: First submitted 2019-01-29; First posted 2019-03-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer; PSA; MRI
Keywords: Prostate cancer; PSA; MRI; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI pathway: Plain biparametric MRI prostate applied to men with elevated PSA, on top of standard screening pathway using PSA and Prostate Health Index
  Interventions: Diagnostic Test: MRI prostate
- Standard screening pathway: Intervention: Using blood tests PSA and Prostate Health Index to screen men at risk of prostate cancer

INTERVENTIONS:
Diagnostic Test: MRI prostate — plain biparametric MRI prostate
  Groups: MRI pathway

SUMMARY:
Under the prostate cancer screening protocol of the project 'Prevention of Obesity-related Cancers', men with elevated PSA with higher prostate cancer risk (PSA 4-10 ng/mL with high Prostate Health Index (PHI) ≥35, or PSA>10 ng/mL) will be offered a prostate biopsy.

In the current study, we would like to offer all screened men with elevated PSA in the range of 4-50 ng/mL a biparametric non-contrast MRI prostate (screening protocol) for any suspicious lesion in the prostate. If there is MRI lesion seen, additional targeted biopsies can be performed on top of the standard systematic prostate biopsies. It has been shown in a clinical Caucasian cohort that doing MRI-targeted biopsies resulted in improved detection of clinically significant prostate cancer compared with standard systematic biopsies.

In this study investigators would like to investigate the benefits of adding MRI prostate and MRI-targeted biopsy in the diagnostic pathway for prostate cancer in a screened cohort of Chinese men at risk of prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the second most common cancer in the world, and its incidence in the Asia-Pacific region is increasing. While serum prostate specific antigen (PSA) level remains the commonest marker for screening of the disease, its specificity is very low. As a result, many patients with elevated PSA are subjected to transrectal ultrasound guided prostatic biopsy (TRUSPB) with negative result, but at the same time faced the complications of bleeding and infection from TRUSPB. Performing a standard 10-12 core systematic prostate biopsy in all men with elevated PSA was shown to miss some clinically significant prostate cancers while over-diagnosing some insignificant prostate cancers. In the European randomized study of screening for prostate cancer (ERSPC), PSA-based screening have resulted in reduced prostate cancer-specific death and metastasis, but there were problems like over-biopsy and over-diagnosis of indolent prostate cancers. The number needed to screen (NNS) to prevent one prostate cancer death was quite high at 781. Therefore, population-wide screening of men with PSA is not commonly applied in most places.

The blood test Prostate Health Index (PHI) provides much better prostate cancer risk stratification than PSA by dividing men with PSA 4-10 ng/mL. Using PHI 35 as a cutoff, clinically significant prostate cancer (any Gleason pattern ≥ 4) was found in only 0.7% in PHI<35, but up to 8.6% in PHI ≥35, a 12 fold difference. The use of PHI test could significantly reduce unnecessary prostate biopsies and was approved by FDA in 2012. Since 2016, the PHI blood test was available in the public health system in Hong Kong for men with PSA 4-10 ng/mL. According to local audit on 2795 men receiving PHI test, about 80% prostate biopsies was avoided. This also resulted in a higher positive biopsy rate (from 10.7% to 26.2%), with the potential of delayed diagnosis in only a minimal proportion of men (0.7%). Currently, PHI is being ordered regularly by Urologists in the public system of Hong Kong for men with PSA 4-10 ng/mL.

In a landmark study by Ahmed et al in 2017, performing multi-parametric MRI prostate before an initial prostate biopsy in a clinical Caucasian cohort has been shown to improve diagnosis of significant prostate cancer by 18%, while reduce diagnosis of insignificant prostate cancer by 5%.

Another Caucasian study by Alberts et al in 2017 in men who undergone the 5th round of screening in European Randomized Study of Screening for Prostate cancer Rotterdam, adding MRI prostate could avoid 65% biopsies and 68% insignificant prostate cancer, while detecting an equal percentage of significant cancers. The role of MRI in an Asian cohort under a screening protocol has not been reported before.

Prostate cancer incidence in Asian is only about one-third of that in Caucasian, and cancer detection rates in different PSA ranges are also 50% less. Reported Caucasian prostate cancer detection rates was 25-50% in men with PSA 4-10 ng/mL and >50% in men with PSA 10-20 ng/mL. In Hong Kong Chinese men, only 15% men with PSA 4-10 ng/mL and 20-30% men with PSA 10-20 ng/mL has prostate cancer. Therefore, screening tools like PHI or MRI are potentially more useful in reducing unnecessary biopsies in Chinese men even in higher PSA ranges (e.g. PSA > 10 ng/mL) due to much lower cancer detection rate.

A multiparametric MRI prostate combines T2-weighted (T2W), Diffusion-weighted imaging (DWI), and Dynamic contrast enhanced (DCE) sequences to aid identification of suspicious malignant lesions in the prostate using a standardized Prostate Imaging - Reporting and Data System (PI-RADS).

In a recently published meta-analysis, it is suggested that a bi-parametric (using only T2W and DWI sequences without contrast) MRI prostate has similar performance compared with a multi-parametric MRI prostate. Omitting the DCE and contrast injection reduces scanning time by 30-50% (down to 15-20 minutes per patient) and avoids risk of gadolinium contrast, especially in men with impaired renal function.

Under the prostate cancer screening protocol of the project 'Prevention of Obesity-related Cancers', men with elevated PSA with higher prostate cancer risk (PSA 4-10 ng/mL with high Prostate Health Index (PHI) ≥35, or PSA>10 ng/mL) will be offered a prostate biopsy.

In the current study, investigators would like to offer all screened men with elevated PSA in the range of 4-50 ng/mL a biparametric non-contrast MRI prostate (screening protocol) for any suspicious lesion in the prostate. If there is MRI lesion seen, additional targeted biopsies can be performed on top of the standard systematic prostate biopsies. It has been shown in a clinical Caucasian cohort that doing MRI-targeted biopsies resulted in improved detection of clinically significant prostate cancer compared with standard systematic biopsies.

In this study investigators would like to investigate the benefits of adding MRI prostate and MRI-targeted biopsy in the diagnostic pathway for prostate cancer in a screened cohort of Chinese men at risk of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Men being screened for prostate cancer in the project 'Prevention of Obesity-related Cancers'
2. Age 50-75
3. Screening naïve, defined as no blood taking for PSA within past 5 years AND no prostate biopsy within past 5 years
4. PSA 4-50 ng/mL
5. Agree for non-contrast MRI scanning of prostate

Exclusion Criteria:

1. Men who are contraindicated for MRI( Pacemaker in-situ, Metallic implants which are not MRI-compatible, or Claustrophobia)
2. Prior history of prostate cancer

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited form the the project 'Prevention of Obesity-related Cancers". 5000 Chinese men between age 50 and 75 will be screened for prostate cancer with the blood test PSA.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
In men with higher risk of prostate cancer, the proportion of men diagnosed with clinically significant prostate cancers on MRI pathway compared with standard screening pathway. | Baseline (only one-time point)
  In men with higher risk of prostate cancer (PSA 10-50 ng/mL, or PSA 4-10 AND Prostate Health Index ≥35), the proportion of men diagnosed with clinically significant prostate cancers on MRI pathway compared with standard screening pathway.
In men with lower risk of prostate cancer the proportion of men diagnosed with clinically significant prostate cancers on MRI pathway compared with standard screening pathway. | Baseline (only one-time point)
  In men with lower risk of prostate cancer (PSA 4-10 ng/mL AND Prostate Health Index <35), the proportion of men diagnosed with clinically significant prostate cancers on MRI pathway compared with standard screening pathway.

SECONDARY OUTCOMES:
Gleason ≥4 cancer AND Maximal cancer core length ≥6mm | Baseline (only one-time point)
  The proportion of men diagnosed with Gleason ≥4 cancer AND Maximal cancer core length ≥6mm
The number of MRI needed to detect one extra clinically significant prostate cancer compared to standard screening pathway | Baseline (only one-time point)
  The number of MRI needed to detect one extra clinically significant prostate
The proportion of men that a biopsy can be avoided by using MRI in higher and lower risk groups | Baseline (only one-time point)
  The proportion of men that a biopsy can be avoided by using MRI in higher and lower risk groups
In men with MRI suspicious lesion (PI-RADS 3 or above), clinically significant prostate cancer diagnosed on Systematic biopsy cores versus targeted biopsy cores | Baseline (only one-time point)
  In men with MRI suspicious lesion (PI-RADS 3 or above), clinically significant prostate cancer diagnosed on Systematic biopsy cores versus targeted biopsy cores

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, FRCP, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - North District Hospital, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu Y, Wang HK, Qu YY, Ye DW. Prostate cancer in East Asia: evolving trend over the last decade. Asian J Androl. 2015 Jan-Feb;17(1):48-57. doi: 10.4103/1008-682X.132780. PMID 25080928
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Berenguer A, Maattanen L, Bangma CH, Aus G, Villers A, Rebillard X, van der Kwast T, Blijenberg BG, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Screening and prostate-cancer mortality in a randomized European study. N Engl J Med. 2009 Mar 26;360(13):1320-8. doi: 10.1056/NEJMoa0810084. Epub 2009 Mar 18. PMID 19297566
- [Background] Braillon A, Dubois G. Re: Fritz H. Schroder, Jonas Hugosson, Sigrid Carlsson, et al. Screening for prostate cancer decreases the risk of developing metastatic disease: findings from the European Randomized Study of Screening for Prostate Cancer (ERSPC). Eur urol 2012;62:745-52. Eur Urol. 2012 Nov;62(5):e89; author reply e90-1. doi: 10.1016/j.eururo.2012.07.031. Epub 2012 Jul 25. No abstract available. PMID 22858456
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Zappa M, Nelen V, Kwiatkowski M, Lujan M, Maattanen L, Lilja H, Denis LJ, Recker F, Paez A, Bangma CH, Carlsson S, Puliti D, Villers A, Rebillard X, Hakama M, Stenman UH, Kujala P, Taari K, Aus G, Huber A, van der Kwast TH, van Schaik RH, de Koning HJ, Moss SM, Auvinen A; ERSPC Investigators. Screening and prostate cancer mortality: results of the European Randomised Study of Screening for Prostate Cancer (ERSPC) at 13 years of follow-up. Lancet. 2014 Dec 6;384(9959):2027-35. doi: 10.1016/S0140-6736(14)60525-0. Epub 2014 Aug 6. PMID 25108889
- [Background] Chiu PK, Roobol MJ, Teoh JY, Lee WM, Yip SY, Hou SM, Bangma CH, Ng CF. Prostate health index (PHI) and prostate-specific antigen (PSA) predictive models for prostate cancer in the Chinese population and the role of digital rectal examination-estimated prostate volume. Int Urol Nephrol. 2016 Oct;48(10):1631-7. doi: 10.1007/s11255-016-1350-8. Epub 2016 Jun 27. PMID 27349564
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Alberts AR, Roobol MJ, Verbeek JFM, Schoots IG, Chiu PK, Osses DF, Tijsterman JD, Beerlage HP, Mannaerts CK, Schimmoller L, Albers P, Arsov C. Prediction of High-grade Prostate Cancer Following Multiparametric Magnetic Resonance Imaging: Improving the Rotterdam European Randomized Study of Screening for Prostate Cancer Risk Calculators. Eur Urol. 2019 Feb;75(2):310-318. doi: 10.1016/j.eururo.2018.07.031. Epub 2018 Aug 3. PMID 30082150
- [Background] Vickers AJ, Cronin AM, Roobol MJ, Hugosson J, Jones JS, Kattan MW, Klein E, Hamdy F, Neal D, Donovan J, Parekh DJ, Ankerst D, Bartsch G, Klocker H, Horninger W, Benchikh A, Salama G, Villers A, Freedland SJ, Moreira DM, Schroder FH, Lilja H. The relationship between prostate-specific antigen and prostate cancer risk: the Prostate Biopsy Collaborative Group. Clin Cancer Res. 2010 Sep 1;16(17):4374-81. doi: 10.1158/1078-0432.CCR-10-1328. Epub 2010 Aug 24. PMID 20736330
- [Background] Chiu PK, Teoh JY, Lee WM, Yee CH, Chan ES, Hou SM, Ng CF. Extended use of Prostate Health Index and percentage of [-2]pro-prostate-specific antigen in Chinese men with prostate specific antigen 10-20 ng/mL and normal digital rectal examination. Investig Clin Urol. 2016 Sep;57(5):336-42. doi: 10.4111/icu.2016.57.5.336. Epub 2016 Aug 31. PMID 27617315
- [Background] Chen R, Ren S; Chinese Prostate Cancer Consortium; Yiu MK, Fai NC, Cheng WS, Ian LH, Naito S, Matsuda T, Kehinde E, Kural A, Chiu JY, Umbas R, Wei Q, Shi X, Zhou L, Huang J, Huang Y, Xie L, Ma L, Yin C, Xu D, Xu K, Ye Z, Liu C, Ye D, Gao X, Fu Q, Hou J, Yuan J, He D, Pan T, Ding Q, Jin F, Shi B, Wang G, Liu X, Wang D, Shen Z, Kong X, Xu W, Deng Y, Xia H, Cohen AN, Gao X, Xu C, Sun Y. Prostate cancer in Asia: A collaborative report. Asian J Urol. 2014 Oct;1(1):15-29. doi: 10.1016/j.ajur.2014.08.007. Epub 2015 Apr 16. PMID 29511634
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH, Moon MH. Head-to-Head Comparison Between Biparametric and Multiparametric MRI for the Diagnosis of Prostate Cancer: A Systematic Review and Meta-Analysis. AJR Am J Roentgenol. 2018 Nov;211(5):W226-W241. doi: 10.2214/AJR.18.19880. Epub 2018 Sep 21. PMID 30240296